CLINICAL TRIAL: NCT06210360
Title: NALIRIFOX as Perioperative Treatment in Patients With High-risk Resectable Pancreatic Cancer : a Multicenter, Randomized, Open-label Trial
Brief Title: Perioperative Treatment in High-risk Resectable Pancreatic Cancer With NALIRIFOX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-PC-03
Record Dates: First submitted 2024-01-02; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Cancer
Keywords: high-risk resectable; NALIRIFOX; perioperative
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: NALIRIFOX + surgery + NALIRIFOX (Experimental): Patients receive 8 cycles of NALIRIFOX. Then undergo surgery and receive 4 cycles of NALIRIFOX after surgery. NALIRIFOX consists of irinotecan liposome injection, oxaliplatin, 5 FU/LV
  Interventions: Drug: Irinotecan liposome injection; Drug: Oxaliplatin; Drug: 5-FU; Drug: LV
- Group B: surgery + NALIRIFOX (Active Comparator): Patients receive 12 cycles of NALIRIFOX after surgery. NALIRIFOX consists of irinotecan liposome injection, oxaliplatin, 5 FU/LV.
  Interventions: Drug: Irinotecan liposome injection; Drug: Oxaliplatin; Drug: 5-FU; Drug: LV

INTERVENTIONS:
Drug: Irinotecan liposome injection — 50 mg/m² on Day 1 of a 14 day cycle
  Other Names: Nal-IRI
Drug: Oxaliplatin — 60 mg/m² on Day 1 of a 14 day cycle
  Other Names: Eloxatin®
Drug: 5-FU — 2400 mg/m² continuous IV infusion in 46 h
  Other Names: 5-Fluorouracil; flurouracil; Adrucil®
Drug: LV — 400 mg/m² on Day 1 of a 14 day cycle
  Other Names: Folinic Acid; Leucovorin

SUMMARY:
This multicentric randomized trial will compare the efficacy and safety of neoadjuvant chemotherapy + surgery + adjuvant chemotherapy or surgery + adjuvant chemotherapy in patients with high-risk resectable pancreatic cancer. NALIRIFOX (5-fluorouracil, leucovorin, irinotecan liposome injection and oxaliplatin) will be used as the chemotherapy regimen.

DETAILED DESCRIPTION:
Liposomal irinotecan is a new pharmaceutical form of traditional irinotecan. It adopts a special loading technology to encapsulate traditional irinotecan in liposomes, which can avoid its hydrolysis under physiological conditions, increase the affinity with cancer cells, overcome drug resistance, increase the drug uptake by cancer cells, reduce the drug dose,improve the efficacy and reduce the toxic side effects. The aim of this study is to compare the efficacy and safety of NALIRIFOX + surgery + NALIRIFOX or surgery + NALIRIFOX in high-risk patients with resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old.
2. Histologically or cytologically proven pancreatic ductal adenocarcinoma.
3. Multidisciplinary assessment as high-risk resectable disease.
4. At least one measurable lesion (according to RECIST v1.1).
5. No prior antitumor therapy for pancreatic cancer.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 ~ 1.
7. The expected survival time ≥3 months.
8. Subject has adequate biological parameters as demonstrated by the following blood counts:

   Absolute neutrophil count (ANC) ≥1.5×10^9/L Platelet count ≥100×10^9/L Hemoglobin (Hgb) ≥90 g/L White blood cell（WBC）≥3.0×10^9/L
9. Adequate hepatic function as evidenced by:

   Serum total bilirubin ≤1.5 × upper limit of normal (ULN), Aspartate aminotransferase (AST) 、alkaline phosphatase（ALP）and alanine aminotransferase (ALT) ≤2.5 × ULN
10. Adequate renal function as evidenced by serum creatinine (Cr)≤1.5 × ULN or creatinine clearance ≥60 mL/min.
11. Agree and be able to comply with the plan during the study period. Provide written informed consent before entering the study screening.

Exclusion Criteria:

1. Any other malignancy within 5 years prior to randomization, with the exception of cured in-situ carcinoma or basal cell carcinoma.
2. Patients with distant metastases and/or can not complete resection.
3. Active, uncontrolled bacterial, viral, or fungal infections that require systemic treatment.
4. Active HIV, HBV, HCV infection.
5. Combined with uncontrollable systemic diseases (such as unstable angina, myocardial infarction, congestive heart failure, severe unstable ventricular arrhythmia, severe pericardial disease history and other cardiovascular diseases; hypertension > grade 2 after medication [CTCAE v5.0], diabetes, etc.)
6. Presence of severe gastrointestinal disease (including active bleeding, > grade 1 obstruction [CTCAE v5.0], or > grade 1 diarrhea [CTCAE v5.0])
7. History of allergy or hypersensitivity to drug or any of their excipients.
8. Patients who have chemotherapy and surgery contraindications.
9. Documented serum albumin ≤3 g/dL
10. Use of strong inhibitors or inducers of CYP3A, CYP2C8 and UGT1A1.
11. Pregnant or breastfeeding women, or subjects of childbearing age who refuse contraception.
12. Participated in other trial within 30 days prior to the first dose of study treatment.
13. Patients who are not suitable to participate in this trial for any reason judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
2-year Overall Survival Rate | 2 years
  Defined as the percentage of patients who are alive at 2 years after randomization (proportion of patients alive will estimated by the survival curve)

SECONDARY OUTCOMES:
Objective Response Rate | 4 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1
Surgical Conversion Rate（R0 / R1 resection） | 5 months
  Defined as the percentage of patients that underwent a R0/R1 resection
R0 resection rate | 5 months
  Defined as the proportion of patients who have achieved R0 resection
Event-free Survival | 1 year
  Defined as the time between signing the informed consent form to the first documentation of event where events considered are 1) disease progression (local recurrence, new lesions or distant metastasis), 2) a second malignant tumor occurs, or 3) death due to any cause
Overall survival | 2 years
  Defined as the time between signing the informed consent form and death due to various causes
Incidence of adverse events | 7 months
  Use NCI-CTCAE version 5.0 for classification and grading

CONTACTS AND LOCATIONS:
Overall Officials: Jin Gang, Professor, Principal Investigator — Changhai Hospital

IPD SHARING:
Plan to Share IPD: No